CLINICAL TRIAL: NCT04252859
Title: [18F]Fluoroestradiol-Positron Emission Tomography (PET)/CT Imaging of Invasive Lobular Carcinoma
Brief Title: [18F]Fluoroestradiol-PET/CT Imaging of Invasive Lobular Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI is leaving the institution.
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HCI128055
Record Dates: First submitted 2020-01-24; First posted 2020-02-05 (Actual); Results first posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-04

CONDITIONS: Invasive Lobular Breast Carcinoma
MeSH Terms: conditions — Carcinoma, Lobular | interventions — proto-oncogene protein c-fes-fps; Fluorine-18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pilot Phase (Experimental): Subjects with biopsy-proven invasive lobular carcinoma (ILC), diagnosed within 12 weeks of imaging, confirmed from biopsy of primary tumor or metastasis, will undergo one Fluorine-18 (18F) -Fluoroestradiol (FES) positron emission tomography/computed tomography (PET/CT) scan and one optional 18F-fluorodeoxyglucose (FDG) PET/CT(if a standard of care scan not already performed).
  For the FES scan, patients are administered a dose of approximately 6 millicurie (mCi) and imaged approximately 60 minutes after injection.
  For the FDG scan, patients are administered a dose of approximately 15 mCi and imaged approximately 60 minutes after injection.
  Interventions: Drug: [18F]Fluoroestradiol (FES) PET/CT
- Expansion Phase (Experimental): Subjects with histologically confirmed estrogen receptor positive (ER+) invasive lobular carcinoma (ILC), diagnosed within 16 weeks of imaging, confirmed from biopsy of primary tumor or metastasis, will undergo one 18F-Fluoroestradiol (FES) PET/CT scan, one optional 18F-FDG PET/CT (if a standard of care scan not already performed), and one optional follow-up FES-PET/CT.
  For the FES scan, patients are administered a dose of approximately 6 mCi and imaged approximately 60 minutes after injection.
  For the FDG scan, patients are administered a dose of approximately 15 mCi and imaged approximately 60 minutes after injection.
  Interventions: Drug: [18F]Fluoroestradiol (FES) PET/CT

INTERVENTIONS:
Drug: [18F]Fluoroestradiol (FES) PET/CT — [18F]Fluoroestradiol (FES) PET/CT for invasive lobular carcinoma (ILC)
  Other Names: Fluorine-18 (18F) Fluoroestradiol

SUMMARY:
FES PET/CT imaging for invasive lobular cancer

DETAILED DESCRIPTION:
According to the National Comprehensive Cancer Network (NCCN) 2018 guidelines 18F-2-fluoro-2-deoxy-D-glucose (FDG)-Positron Emission Tomography/Computed Tomography (PET/CT) may be performed as an alternative to a contrast-enhanced CT of the chest, abdomen and pelvis and Tc-99m methylene diphosphonate (MDP) bone scan for evaluation of distant metastatic disease in newly diagnosed stage III breast cancer patients. FDG-PET/CT is usually not obtained for stage I or stage II breast cancer patients as change in patient management is rare. Prior studies have demonstrated FDG-PET/CT can identify sites of unsuspected metastatic disease in newly diagnosed breast cancer patients thereby altering treatment decisions given that palliative management is typical for stage IV disease, whereas neoadjuvant therapy followed by surgery and postoperative radiation may be considered for stage II and operable stage III disease. These guidelines consider invasive breast cancer as a single entity and do not consider whether tailoring imaging techniques for subtypes of breast cancer may be beneficial. However, prior research suggests that FDG-PET/CT may be more appropriate as an alternative to CT and bone scan for patients with invasive ductal carcinoma (IDC) rather than invasive lobular carcinoma (ILC) as FDG demonstrates comparatively reduced sensitivity for ILC metastases. Compared to IDC, ILC is more often occult on mammography, ultrasound, and FDG-PET/CT; which is of importance for clinical management as ILC is more often multifocal and bilateral compared to IDC. Clinical breast examination also has lower sensitivity for detection of ILC compared to IDC, even for large tumors, as ILC may be indistinguishable from normal breast tissue on palpation.

A prior study evaluating systemic staging of newly diagnosed patients with stage I-III invasive breast cancer found that FDG-PET/CT is 1.98 times less likely to reveal unsuspected distant metastatic disease for women with ILC compared to IDC. In this study, all IDC metastases demonstrated FDG avidity whereas 25% of ILC metastases (3 of 12) were not FDG avid. Detection of local axillary metastatic disease on FDG-PET/CT was also lower for ILC (0 of 146 patients) compared to IDC (7 of 89 patients) despite data from the Surveillance, Epidemiology and End Results (SEER) database demonstrating similar rates for lymph node metastases between IDC and ILC. Another study evaluating FDG-PET/CT for the diagnosis of primary breast cancer found that the false negative rate for detection of ILC by FDG was 65% (15 of 23 cases) compared to 23% for IDC (23 of 97 cases) when matching for tumors of the same size. A final study reported a false negative rate of FDG for ILC detection of 13% (2 of 15 patients). Mechanistically, ILC may not take up FDG as avidly as IDC due to lower tumor microvascularity, cellular density, proliferation rate, and number of glucose transporters (GLUT). ILC osseous metastatic disease is also more frequently occult on FDG-PET/CT compared to IDC as ILC osseous metastases are more frequently sclerotic, whereas FDG-PET/CT is more sensitive for lytic osseous metastases. Sclerotic ILC osseous metastases also may be indistinguishable from benign bone islands on CT at initial staging, thereby necessitating biopsy or imaging follow-up for confirmation of osseous metastatic disease. Improved imaging strategies for primary and metastatic ILC are therefore warranted.

Multiple studies have proven the efficacy of FES-PET/CT for imaging evaluation of ER+ invasive breast malignancy (evaluating both IDC and ILC together, with the large majority of cases comprising IDC) but, to our knowledge, no prior study has focused FES-PET/CT evaluation only to cases of ILC, nor have prior studies compared FES-PET/CT directly with FDG-PET/CT for evaluation of newly diagnosed ILC. Given that all prior studies on FES-PET/CT have grouped a small number of ILC cases with a larger number of IDC cases, the imaging performance of FES-PET/CT specifically for ILC is unknown. ILC demonstrates higher rates of ER positivity than IDC with prior studies showing greater than 90% positivity for cases of ILC. Data from the SEER database also shows ILC demonstrates higher overall expression of ER than IDC (ILC 95% positive for ER, n=17,503 vs IDC 74% positive for ER, n=172,379). FES-PET/CT may therefore be suitable for imaging evaluation of a high proportion of patients with ILC.

ELIGIBILITY:
FOR PILOT PHASE COMPLETED IN 2021:

Inclusion Criteria:

* Adults aged 18 years or greater
* All patients or legal guardians are willing and able to sign a written informed consent and HIPAA authorization in accordance with local and institutional guidelines.
* Histologically confirmed invasive lobular carcinoma within the past 12 weeks confirmed from biopsy of primary tumor or metastasis.
* Patient is willing to have their clinical records reviewed for at least 24 months after enrollment.

FOR PILOT PHASE COMPLETED IN 2021:

Exclusion Criteria:

* Patients with known allergic or hypersensitivity reactions to previously administered radiopharmaceuticals. Patients with significant drug or other allergies or autoimmune diseases may be enrolled at the Investigator's discretion.
* Patients who require monitored anesthesia for PET/CT scanning.
* Patients who are too claustrophobic to undergo PET/CT scanning.
* Pregnancy or current breast feeding.
* Any patient that is medically unstable defined as patient requiring inpatient hospitalization or needing evaluation at an acute care or urgent care facility at time of imaging.
* Patients undergoing treatment with estrogen receptor agonists (such as fulvestrant and tamoxifen) within 5 weeks of the FES-PET/CT scan. (Note that aromatase inhibitors and luteinizing hormone-releasing hormone agonists do not affect ER expression, or binding of FES to ER, and do not need to be discontinued or considered for inclusion or exclusion of patients).
* Patient who have had the site(s) of biopsy proven invasive lobular carcinoma surgically resected.

FOR EXPANSION PHASE ADDED IN MARCH 2022 AMENDMENT:

INCLUSION CRITERIA:

* Adults aged 18 years or greater
* All patients or legal guardians are willing and able to sign a written informed consent and HIPAA authorization in accordance with local and institutional guidelines.
* Patient must qualify for one of the following:

Primary endpoint analysis/Primary Arm:

Histologically confirmed ER+ invasive lobular carcinoma within the past 16 weeks confirmed from biopsy of primary tumor or metastasis (n=40).

Exploratory Arm 1:

Histologically confirmed ER+ invasive lobular carcinoma at any time in the past, confirmed from biopsy of primary tumor or metastasis, with confirmed or imaging suspected metastatic disease, currently on antihormonal therapy or chemotherapy (n=10).

Exploratory Arm 2:

Histologically confirmed ER- invasive lobular carcinoma (at any point) at any site with biopsy-proven or imaging suspected metastatic ILC (n=5).

* Patient is willing to have their clinical records reviewed, and be contacted by phone during follow-up intervals specified, for approximately 60 months after enrollment.
* Patient is willing to provide baseline blood specimens for circulating tumor DNA (ctDNA) analysis.

FOR EXPANSION PHASE ADDED IN MARCH 2022 AMENDMENT:

EXCLUSION CRITERIA:

* Patients with known allergic or hypersensitivity reactions to previously administered radiopharmaceuticals. Patients with significant drug or other allergies or autoimmune diseases may be enrolled at the Investigator's discretion.
* Patients who require monitored anesthesia for PET/CT scanning.
* Patients who are too claustrophobic to undergo PET/CT scanning.
* Pregnancy or current breast feeding.
* Patient who have had the site(s) of biopsy proven invasive lobular carcinoma surgically resected. Note: This does not apply for participants being enrolled for Exploratory Arm 1.
* Patients undergoing treatment with estrogen receptor agonists (such as fulvestrant and tamoxifen) within 5 weeks of the FES-PET/CT scan.

(Note that aromatase inhibitors and luteinizing hormone-releasing hormone agonists do not affect ER expression, or binding of FES to ER, and do not need to be discontinued or considered for inclusion or exclusion of patients). Note: This does not apply for participants being enrolled for Exploratory Arm 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2020-12-11 (Actual); Primary Completion 2024-12-07 (Actual); Study Completion 2024-12-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Yap, PhD, Principal Investigator — Huntsman Cancer Institute/ University of Utah
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Covington MF, Hoffman JM, Morton KA, Buckway B, Boucher KM, Rosenthal RE, Porretta JM, Brownson KE, Matsen CB, Vaklavas C, Ward JH, Wei M, Buys SS, Chittoria N, Yakish ED, Archibald ZG, Burrell LD, Butterfield RI, Yap JT. Prospective Pilot Study of 18F-Fluoroestradiol PET/CT in Patients With Invasive Lobular Carcinomas. AJR Am J Roentgenol. 2023 Aug;221(2):228-239. doi: 10.2214/AJR.22.28809. Epub 2023 Mar 15. PMID 36919879

RESULTS

PARTICIPANT FLOW:
Groups:
- Pilot Phase: Subjects with biopsy-proven invasive lobular carcinoma (ILC), diagnosed within 12 weeks of imaging, will undergo one Fluorine-18 (18F) -Fluoroestradiol (FES) positron emission tomography/computed tomography (PET/CT) scan and one optional 18F-fluorodeoxyglucose (FDG) PET/CT(if a standard of care scan not already performed).
  For the FES scan, patients are administered a dose of approximately 6 millicurie (mCi) and imaged approximately 60 minutes after injection.
  For the FDG scan, patients are administered a dose of approximately 15 mCi and imaged approximately 60 minutes after injection.
  [18F]Fluoroestradiol (FES) PET/CT: [18F]Fluoroestradiol (FES) PET/CT for invasive lobular carcinoma (ILC)
- Expansion Phase: Subjects with histologically confirmed estrogen receptor positive (ER+) invasive lobular carcinoma (ILC), diagnosed within 16 weeks of imaging, will undergo one 18F-Fluoroestradiol (FES) PET/CT scan, one optional 18F-fluorodeoxyglucose (FDG) PET/CT (if a standard of care scan not already performed), and one optional follow-up FES-PET/CT.
  For the FES scan, patients are administered a dose of approximately 6 mCi and imaged approximately 60 minutes after injection.
  For the FDG scan, patients are administered a dose of approximately 15 mCi and imaged approximately 60 minutes after injection.
  [18F]Fluoroestradiol (FES) PET/CT: [18F]Fluoroestradiol (FES) PET/CT for invasive lobular carcinoma (ILC)
Period: Overall Study
Arm/Group | Pilot Phase | Expansion Phase
Started | 19 | 25
Completed | 19 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Pilot Phase: Subjects with biopsy-proven invasive lobular carcinoma (ILC), diagnosed within 12 weeks of imaging, will undergo one 18F-Fluoroestradiol (FES) PET/CT scan and one optional 18F-FDG PET/CT(if a standard of care scan not already performed).
- Expansion Phase: Subjects with histologically confirmed estrogen receptor positive (ER+) invasive lobular carcinoma (ILC), diagnosed within 16 weeks of imaging, will undergo one 18F-Fluoroestradiol (FES) PET/CT scan, one optional 18F-FDG PET/CT (if a standard of care scan not already performed), and one optional follow-up FES-PET/CT.
- Total: Total of all reporting groups
Arm/Group | Pilot Phase | Expansion Phase | Total
Number analyzed (Participants) | 17 | 25 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 17 | 23
  >=65 years | 11 | 8 | 19
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.6 (13.5) | 61.4 (11.1) | 60.7 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 25 | 42
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 5
  Not Hispanic or Latino | 16 | 21 | 37
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 16 | 21 | 37
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17 | 25 | 42

OUTCOME MEASURES:

1. Primary Outcome: Positive Detection Rate of Invasive Lobular Carcinoma (ILC)
Description: The number of known ILC sites that demonstrate abnormal FES uptake by FES-PET/CT, defined as focal uptake above background with standardized uptake value (SUV) max of 1.5 or greater, relative to the total number of known ILC sites.
Time Frame: At time of baseline FES-PET/CT imaging
Population: This primary endpoint was evaluated using data collected during Pilot Phase only.
Measure: Count of Units; unit: Lesions
Units Other Than Participants: Lesions
Groups:
- Pilot Phase: Subjects with biopsy-proven invasive lobular carcinoma (ILC), diagnosed within 12 weeks of imaging, will undergo one 18F-Fluoroestradiol (FES) PET/CT scan and one optional 18F-FDG PET/CT(if a standard of care scan not already performed).
  For the FES scan, patients are administered a dose of approximately 6 mCi and imaged approximately 60 minutes after injection.
  For the FDG scan, patients are administered a dose of approximately 15 mCi and imaged approximately 60 minutes after injection.
  [18F]Fluoroestradiol (FES) PET/CT: [18F]Fluoroestradiol (FES) PET/CT for invasive lobular carcinoma (ILC)
- Expansion Phase: Subjects with histologically confirmed estrogen receptor positive (ER+) invasive lobular carcinoma (ILC), diagnosed within 16 weeks of imaging, will undergo one 18F-Fluoroestradiol (FES) PET/CT scan, one optional 18F-FDG PET/CT (if a standard of care scan not already performed), and one optional follow-up FES-PET/CT.
  For the FES scan, patients are administered a dose of approximately 6 mCi and imaged approximately 60 minutes after injection.
  For the FDG scan, patients are administered a dose of approximately 15 mCi and imaged approximately 60 minutes after injection.
  [18F]Fluoroestradiol (FES) PET/CT: [18F]Fluoroestradiol (FES) PET/CT for invasive lobular carcinoma (ILC)
Arm/Group | Pilot Phase | Expansion Phase
Number analyzed (Participants) | 17 | 0
Number analyzed (Lesions) | 25 | 0
Lesions | 22 |

2. Primary Outcome: Change in Staging of Patients With Newly Diagnosed ILC
Description: Blinded analysis was performed to determine staging fore each patient using FES-PET/CT imaging only and compared to the clinical stage assigned to each patient using a standard-of-care evaluation.
Time Frame: At time of baseline FES-PET/CT imaging
Population: This primary endpoint was evaluated using data collected during Expansion Phase only.
Measure: Count of Participants; unit: Participants
Groups:
- Pilot Phase: Subjects with biopsy-proven invasive lobular carcinoma (ILC), diagnosed within 12 weeks of imaging, confirmed from biopsy of primary tumor or metastasis, will undergo one 18F-Fluoroestradiol (FES) PET/CT scan and one optional 18F-FDG PET/CT(if a standard of care scan not already performed).
  For the FES scan, patients are administered a dose of approximately 6 mCi and imaged approximately 60 minutes after injection.
  For the FDG scan, patients are administered a dose of approximately 15 mCi and imaged approximately 60 minutes after injection.
  [18F]Fluoroestradiol (FES) PET/CT: [18F]Fluoroestradiol (FES) PET/CT for invasive lobular carcinoma (ILC)
- Expansion Phase: Subjects with histologically confirmed estrogen receptor positive (ER+) invasive lobular carcinoma (ILC), diagnosed within 16 weeks of imaging, confirmed from biopsy of primary tumor or metastasis, will undergo one 18F-Fluoroestradiol (FES) PET/CT scan, one optional 18F-FDG PET/CT (if a standard of care scan not already performed), and one optional follow-up FES-PET/CT.
  For the FES scan, patients are administered a dose of approximately 6 mCi and imaged approximately 60 minutes after injection.
  For the FDG scan, patients are administered a dose of approximately 15 mCi and imaged approximately 60 minutes after injection.
  [18F]Fluoroestradiol (FES) PET/CT: [18F]Fluoroestradiol (FES) PET/CT for invasive lobular carcinoma (ILC)
Arm/Group | Pilot Phase | Expansion Phase
Number analyzed (Participants) | 0 | 25
Participants |  | 9

3. Secondary Outcome: Rate of Estrogen Receptor Positive (ER+) ILC That Does Not Demonstrate Positive FES Uptake
Description: The number of known ER+ ILC sites that do not demonstrate abnormal FES uptake by FES-PET/CT, defined as focal uptake above background with SUV max of 1.5 or greater, relative to the total number of known ER+ ILC sites.
Time Frame: At time of baseline FES-PET/CT imaging
Population: This secondary endpoint was evaluated using data collected during Pilot Phase only.
Measure: Count of Units; unit: Lesions
Units Other Than Participants: Lesions
Arm/Group | Pilot Phase | Expansion Phase
Number analyzed (Participants) | 17 | 0
Number analyzed (Lesions) | 20 | 0
Lesions | 3 |

4. Secondary Outcome: Rate of Estrogen Receptor Negative (ER-) ILC That Does Demonstrate Positive FES Uptake
Description: The number of known ER- ILC sites that demonstrate abnormal FES uptake by FES-PET/CT, defined as focal uptake above background with SUV max of 1.5 or greater, relative to the total number of known ER- ILC sites.
Time Frame: This secondary endpoint was evaluated using data collected during Pilot Phase only.
Population: This secondary endpoint was evaluated using data collected during Pilot Phase only.
Measure: Count of Units; unit: Lesion
Units Other Than Participants: Lesion
Arm/Group | Pilot Phase | Expansion Phase
Number analyzed (Participants) | 17 | 0
Number analyzed (Lesion) | 1 | 0
Lesion | 1 |

5. Secondary Outcome: Rate of Same-patient (Inter-tumoral) Heterogeneous FES Uptake
Description: Number of patients demonstrating a presence of FES uptake with SUV max of 1.5 or greater in some but not all biopsy proven or suspected metastatic lesions.
Time Frame: At time of baseline FES-PET/CT imaging
Population: This secondary endpoint was evaluated using data collected during Pilot Phase only.
Measure: Count of Participants; unit: Participants
Arm/Group | Pilot Phase | Expansion Phase
Number analyzed (Participants) | 17 | 0
Participants | 1 |

6. Secondary Outcome: Rate of Discordant Uptake (FES Positive/FDG Negative or FES Negative/FDG Positive)
Description: Differences between FDG- and FES uptake. Discordant uptake will be evaluated for any histologically confirmed site of ILC before or after enrollment. Only lesions in patients who underwent both FES- and FDG-PET/CT scans will be included in this assessment.
  Discordant uptake is defined as individual lesions that show either positive FES uptake and negative FDG uptake, or negative FES uptake and positive FDG uptake.
Time Frame: At time of baseline FES-PET/CT imaging and FDG-PET/CT (done within four weeks of FES-PET/CT imaging)
Population: This secondary endpoint was evaluated using data collected during Pilot Phase only.
Measure: Count of Units; unit: Lesions
Units Other Than Participants: Lesions
Arm/Group | Pilot Phase | Expansion Phase
Number analyzed (Participants) | 13 | 0
Number analyzed (Lesions) | 23 | 0
Lesions
  FES positive/FDG negative | 4 |
  FES negative/FDG positive | 1 |
  FES postive/FDG positive | 16 |
  FES negative/FDG negative | 2 |

7. Secondary Outcome: Correlation of Lesion Uptake Between FES and FDG.
Description: SUVmax values are compared for FES- and FDG-PET/CT within sites of abnormal uptake.
Time Frame: At time of baseline FES-PET/CT imaging and FDG-PET/CT (done within four weeks of FES-PET/CT imaging)
Population: This outcome measure is not applicable for the expansion phase.
Measure: Mean (95% Confidence Interval); unit: Lesions
Units Other Than Participants: Lesions
Arm/Group | Pilot Phase | Expansion Phase
Number analyzed (Participants) | 19 | 0
Number analyzed (Lesions) | 19 | 0
Lesions
  FES Treated Lesions | 3.79 [2.51 to 6.30] |
  FDG-PET/CT Treated Lesions | 3.97 [2.62 to 6.59] |

8. Secondary Outcome: Ability to Predict Patient Stage at Presentation by Quantity of Methylated ctDNA at Baseline
Description: This outcome measure will assess whether the quantity of methylated ctDNA at baseline predicts patient stage at presentation per the American Joint Committee on Cancer (AJCC) TNM system. Spearman correlation would be used to assess the correlation between circulating tumor DNA (ctDNA) and stage.
  This outcome measure can not be reported as technical issues prevented the ctDNA analysis.
Time Frame: At time of baseline FES-PET/CT imaging
Population: This endpoint could not be evaluated due to technical issues encountered during ctDNA analysis.
Arm/Group | Pilot Phase | Expansion Phase
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Assess Correlation Between Methylated ctDNA and Overall Survival
Description: To assess whether quantity of methylated ctDNA at baseline predicts survival at each follow-up interval starting at 6 months (follow-up performed at 6, 12, 18, 24, 36, 48 and 60 months). A proportional hazards model will be used to assess the relationship between methylated ctDNA and overall survival. To determine the relationship at various time points, the analysis will be performed with censoring at 6, 12, 18, 24, 36, 48 and 60 months.
  This outcome measure can not be reported as technical issues prevented the ctDNA analysis.
Time Frame: ctDNA samples collected for all patients at baseline and collected at 6, 12, 18, 24, 36, 48, and 60 months after baseline for patients who consented to additional collection
Population: This endpoint could not be evaluated due to technical issues encountered during ctDNA analysis.
Arm/Group | Pilot Phase | Expansion Phase
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Relationship Between Presence of Heterogeneous FES-PET/CT Uptake at Baseline and Overall Survival
Description: To assess whether heterogeneous FES-PET/CT uptake at baseline (yes/no), defined as abnormal FES uptake in some but not all proven or suspected ILC lesions, predicts survival at each follow-up interval starting at 6 months (follow-up performed at 6, 12, 18 months).
  Due to early termination of the study, subject are censored at the end of study date. No participants had heterogeneous FES-PET/CT uptake at baseline. No participants died on study.
Time Frame: Survival is assessed from baseline to study closure (up to 27 months from baseline FES-PET/CT)
Population: Only three participants were evaluable for this endpoint, none had heterogeneous FES-PET/CT uptake at baseline.
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Pilot Phase | Expansion Phase
Number analyzed (Participants) | 0 | 3
months |  | 25.5 [21.67 to 46.82]

ADVERSE EVENTS:
Time Frame: Adverse events and Serious Adverse Events were followed while the subjects were on the study; up to 3 days from initiation of the study intervention. Due to early termination of the study, survival was censored at the study completion date. Survival was followed for up to 27.1 months from baseline.
Arm/Group | Pilot Phase | Expansion Phase
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/25
Other Adverse Events (participants affected / at risk) | 7/17 | 0/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pilot Phase (N=17) | Expansion Phase (N=25)
Diarrhea (Gastrointestinal disorders) | 2 (3) | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | NA
Hypertension (Vascular disorders) | 1 (1) | NA
Nausea (Gastrointestinal disorders) | 2 (2) | NA
Belching (Gastrointestinal disorders) | 1 (1) | NA
Vomiting (Gastrointestinal disorders) | 2 (2) | NA
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) | NA — Mild redness of the skin
Non-cardiac chest pain (General disorders) | 1 (1) | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-12-01): https://cdn.clinicaltrials.gov/large-docs/59/NCT04252859/Prot_SAP_000.pdf
  • Informed Consent Form (2024-06-12): https://cdn.clinicaltrials.gov/large-docs/59/NCT04252859/ICF_001.pdf